CLINICAL TRIAL: NCT06096870
Title: Phase II Trial of Enzalutamide and PDS01ADC in PET Positive Recurrent Prostate Cancer (pprPC) Without Testosterone Lowering Therapy
Brief Title: Enzalutamide and PDS01ADC in PET Positive Recurrent Prostate Cancer (pprPC) Without Testosterone Lowering Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10001556; 001556-C
Record Dates: First submitted 2023-10-21; First posted 2023-10-24 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10-16

CONDITIONS: Prostate Cancer; Recurrent Prostate Cancer; PET Positive
Keywords: Combination Therapy; Recurrent Prostate Cancer; PET Positive; Enzalutamide; PDS01ADC
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Enzalutamide
  Interventions: Drug: Enzalutamide
- Arm 2 (Experimental): Enzalutamide+PDS01ADC
  Interventions: Drug: Enzalutamide; Drug: PDS01ADC

INTERVENTIONS:
Drug: Enzalutamide — Enzalutamide at 160 mg once daily on every day of the cycle (every 28 days)
Drug: PDS01ADC — PDS01ADC at 12.0 microgram/kg by subcutaneous injection (every 28 days)
  Arms: Arm 2

SUMMARY:
Background:

Prostate cancer may return after treatment in 30,000 to 50,000 people each year. There is no clear best way to treat these people. Better treatments are needed.

Objective:

To test a study drug (enzalutamide), both alone and combined with a second drug (PDS01ADC), in people with prostate cancer that returned after treatment.

Eligibility:

People aged 18 years and older with prostate cancer that returned after treatment.

Design:

Participants will be screened. They will have a physical exam, with blood tests. All their urine will be collected for 24 hours. They will have imaging scans of their chest, abdomen, pelvis, and bones. Their ability to perform everyday activities will be assessed. They may opt to give a stool sample.

Participants will be treated in 4-week cycles.

Enzalutamide is a pill taken by mouth once a day, every day. All participants will be given a supply of this drug to take at home.

PDS01ADC is injected under the skin once a month, on the first day of each cycle. Half of the participants will receive both drugs.

All participants will visit the clinic once a month. Each visit should last no more than 8 hours. Blood and urine tests will be repeated.

All participants will receive the study treatment for 3 cycles. Some participants may need 3 more cycles of treatment with enzalutamide only. This re-treatment can be done only once.

Participants will have a follow-up visit 1 month after they finish treatment. After that, they will have visits every 6 weeks for up to 5 years. Imaging scans and blood tests will be repeated.

...

DETAILED DESCRIPTION:
* Enzalutamide given with androgen deprivation therapy (ADT) is Food and Drug Administration (FDA) approved for the treatment of metastatic prostate cancer based on conventional computed tomography (CT) and Tc99 scan.
* Enzalutamide for 3 months (short course) given without ADT has demonstrated the ability to control prostate-specific antigen (PSA) in recurrent prostate cancer for nearly a year, delaying the need for additional therapy.
* Enzalutamide without ADT was very well tolerated in our previous study, a prerequisite for any therapy in recurrent disease where patients may not have symptoms from prostate cancer for 5-10 years.
* Enzalutamide without ADT demonstrated the ability to enhance natural killer (NK) cells and decrease myeloid-derived suppressor cells.
* PDS01ADC is an immunocytokine that binds to areas of necrotic tumors. Preclinical data have demonstrated that PDS01ADC delivery to the tumor is enhanced by cytotoxic therapies such as radiation and chemotherapy.
* PDS01ADC has been shown to be well tolerated and even induce PSA responses in patients with recurrent prostate cancer.
* PDS01ADC has also been able to enhance NK cells in prostate cancer patients.
* Higher levels of NK cells have been associated with better clinical outcomes in prostate cancer.
* Prostate-specific membrane antigen (PSMA) positron emission tomography (PET) imaging is now approved in recurrent prostate cancer. No trial has prospectively evaluated an anti-androgen therapy (e.g., enzalutamide) without ADT in this population. If changes in imaging are seen similar to the PSA responses noted previously, these findings may demonstrate the efficacy of enzalutamide-based regimens in recurrent prostate cancer.
* Given that enzalutamide is cytotoxic and will induce necrosis, there is a rationale to combine it with the necrosis-targeting agent PDS01ADC. The fact that both enhance NK cells, which have been associated with better clinical outcomes adds further rationale to this combination.

Objective:

-To determine if the combination of enzalutamide and immunotherapy (PDS01ADC) is associated with an increase in the duration of PSA suppression compared to that of enzalutamide alone in participants with PET Positive Recurrent Prostate Cancer (pprPC).

Eligibility:

* Participant must provide documentation of histologic or cytological confirmation of prostate cancer or tumor sample for diagnosis confirmation. Note: in the absence of pathology or documentation, participant must have a rising PSA, PSMA plus disease, and his history consistent with prostate cancer as documented by the investigator.
* History of primary treatment for prostate cancer (either surgery or radiation).
* PSA doubling time within less than 1 year before treatment initiation.
* Testosterone >100 ng/dL.
* Age >=18 years.
* Evidence of prostate cancer on PSMA PET/CT scan.
* Negative Tc99 Bone Scan.
* No evidence of soft tissue disease on the CT scan (or MRI) per the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1).

Design:

* This is an open-label phase II clinical trial with two treatment arms: Arm 1 (enzalutamide) and Arm 2 (enzalutamide plus PDS01ADC).
* After enrollment, participants will be randomized between Arms 1 and 2 and receive 3 cycles of treatment of enzalutamide or enzalutamide and PDS01ADC.
* During off treatment monitoring period following the third cycle, participants who experience PSA recovery to baseline will have a second course of enzalutamide treatment only (3 cycles total).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participant must provide documentation of histologic or cytological confirmation of prostate cancer or tumor sample for diagnosis confirmation. Note: in the absence of pathology or documentation, participant must have a rising PSA, PSMA+ disease, and his history consistent with prostate cancer as documented by the investigator.
* History of primary treatment for prostate cancer (either surgery or radiation).
* Prostate-specific antigen (PSA) doubling time within less than 12 months.
* Testosterone >100 ng/dL.
* Age >=18 years.
* Evidence of prostate cancer on PSMA PET/CT scan.
* Eastern Cooperative Oncology Group (ECOG) performance status <2.
* Men must agree to use an effective method of contraception (barrier or surgical sterilization) after study entry and for 3 months after completion of enzalutamide or PDS01ADC therapy whatever comes later.
* Participants must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count (ANC) >=1,500/microliter, without granulocyte colony-stimulating factor (G-CSF) support
  * Platelets >=100,000/microliter
  * Aspartate aminotransferase (AST) /Alanine aminotransferase (ALT) <=2.5 x institutional upper limit of normal (ULN)
  * Hemoglobin (Hgb) >= 10 g/dL (packed red blood cell (pRBC) transfusions are not allowed to achieve acceptable Hgb)
  * Total bilirubin <= 1.5 x ULN, OR <= 3.0 ULN in participants with Gilbert s syndrome
  * Serum albumin >= 2.8 g/dL
  * Creatinine < 1.5 X institution ULN

OR

--Measured or calculated creatinine clearance (CrCl) (estimated glomerular filtration rate (eGFR) may also be used in place of CrCl) > 45 mL/min/1.73 m^2 for participant with creatinine levels > 1.5 x institutional ULN

* Hepatitis B virus (HBV)-infected participants can be enrolled if HBV DNA is undetectable at screening. Hepatitis C virus (HCV)-infected participants can be enrolled if the HCV RNA level is undetectable at screening. Human immunodeficiency virus (HIV)-positive participants can be enrolled if HIV DNA is undetectable.
* Participants must be able to swallow tablets/capsules.
* Participants must be able to understand and willing to sign a written informed consent document.

EXCLUSION CRITERIA:

* Evidence of soft tissue disease on CT scan (or magnetic resonance imaging (MRI) if assessment cannot be done by CT scan) per RECIST 1.1 criteria (lymph nodes up to 2.0 cm in the shortest dimension are allowed).
* Evidence of bone lesions on Tc99 bone scan.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study drugs or imaging agents used in the study.
* Any medical condition that requires chronic systemic steroid therapy, or any other form of immunosuppressive medication (inhaled and topical steroids are permitted).
* History of seizures within the last 10 years.
* Therapy with strong inhibitors or inducers of CYP2C8 or CYP3A4 (https://druginteractions.medicine.iu.edu/MainTable.aspx) within 5 half-lives prior to the study treatment initiation.
* Participants with prior malignancy active within 3 years prior to study treatment initiation except for locally curable cancers that have been apparently cured such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the breast.
* Uncontrolled intercurrent illness that would limit compliance with study requirements.

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine if the combination of enzalutamide and PDS01ADC is associated with an increase in the duration of PSA suppression compared to that of enzalutamide alone | 5 years
  Kaplan-Meier curves and a one-tailed log-rank test. The median time to loss of PSA control on each arm will be reported along with a 95% confidence interval; in addition, based on the result from the prior trial, the probability of PSA control at 224 days (approximately 7 months) will also be reported on both arms, along with 95% confidence intervals

SECONDARY OUTCOMES:
PET changes after enzalutamide with and without PDS01ADC treatment | 1 year
  PET changes will be reported descriptively
Safety of study treatment | until 30 days after last dose of study drug
  Safety will be evaluated by determining the frequency of adverse events among treated participants and reporting the results, by maximum grade of event and type of toxicity noted
Evaluate immune response | 1 year
  Results of peripheral immune cell subsets including CD4 and CD8 T cells, NK cells, Tregs, and MDSCs measurements will be reported descriptively
PSA detection | 1 year
  The proportion of participants with undetectable PSA at 12 months will be reported along with a 95% confidence interval

CONTACTS AND LOCATIONS:
Overall Officials: Ravi A Madan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001556-C.html